CLINICAL TRIAL: NCT04630470
Title: Effect of Massage Therapy With Lavender Oil on Severity of Restless Legs Syndrome and Quality of Life in Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Effect of Massage Therapy on Severity of Restless Legs Syndrome and Quality of Life in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayser DÖNER, Research Assistants, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Interventional
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Hemodialysis
Keywords: Hemodialysis,; restless leg,; lavender oil,; massage,; quality of life
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Massage; lavender oil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The placebo control group (Placebo Comparator): Each patient received the massage therapy with baby oil on both lower leg areas for 10 minutes on each leg, for 4 weeks, three times a week, in the first half of the HD session (first 2 hours).
  Interventions: Behavioral: massage therapy with baby oil
- The study group (Experimental): Each patient received the massage therapy with lavender oil on both lower legs for 10 minutes on each leg, for 4 weeks, three times a week, in the first half of the HD session (first 2 hours).
  Interventions: Behavioral: massage therapy with lavender oil

INTERVENTIONS:
Behavioral: massage therapy with lavender oil — massage therapy with lavender oil-on both lower leg areas, for 10 minutes on each leg, for 4 weeks, three times a week, in the HD sessions
  Arms: The study group
Behavioral: massage therapy with baby oil — massage therapy with baby oil-on both lower leg areas, for 10 minutes on each leg, for 4 weeks, three times a week, in the HD sessions
  Arms: The placebo control group

SUMMARY:
This randomized controlled trial was conducted to determine the effect of the massage, applied with 5% lavender oil for the individuals receiving HD therapy, in the first half of HD session three times a week for four weeks on both legs for 10 minutes in each leg, on severity of RLS and quality of life. The study was completed with 58 patients including 31 people in the intervention group and 27 people in the placebo control group, in 7 hemodialysis centers located in a city center.

DETAILED DESCRIPTION:
The restless leg syndrome (RLS) is among the most common problems for the individuals undergoing hemodialysis (HD) therapy. This randomized controlled trial was conducted to determine the effect of the massage, applied with 5% lavender oil for the individuals receiving HD therapy, in the first half of HD session three times a week for four weeks on both legs for 10 minutes in each leg, on severity of RLS and quality of life. The study was completed with 58 patients including 31 people in the intervention group and 27 people in the placebo control group, in 7 hemodialysis centers located in a city center. The ethics committee approval, informed consent of the individuals and the institutional permission were obtained. The data were collected using the patient information form, RLS Severity Rating Scale, Kidney Disease Quality of Life Questionnaire (KDQOLTM-36) and patient follow-up charts. In accordance with the massage application protocol, those in the intervention group were massaged with lavender oil and those in the placebo group were massaged with baby oil. Chi-square test, t test, repeated measures one-way analysis of variance, and Pearson correlation analysis tests were used to assess the data. In the comparisons, the value of p<0.05 was accepted as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* were not pregnant or did not plan pregnancy
* were diagnosed with RLS by a physician
* had at least mild RLS based on the RLS Severity Rating Scale
* had received HD treatment in the HD units for at least 3 months and three sessions per week
* had continued the dialysis treatment at the same institution
* had not changed the treatment schedule before the massage therapy and throughout the study
* could understand and communicate in Turkish

Exclusion Criteria:

* Patients with an allergy to lavender oil
* had an open wound that would hinder the massage therapy
* had lower leg problems such as neuropathy
* had a neurological disease such as epilepsy, Alzheimer's disease, Parkinson's disease, or multiple sclerosis
* had a history of other CIT methods applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
RLS Severity Rating Scale | change from baseline score at the end of one month
  The RLS Severity Rating Scale was developed in 2003 by the International Restless Legs Syndrome Study Group. The scale was applied in the selection of patients and in the weekly evaluation of RLS severity. The scale comprised ten questions; each question was scored between 0 and 4. Questions 1, 2, 4, 6, 7, and 8 were related to RLS symptoms, questions 5, 9, and 10 were related to the effect of the disease on the mental state and daily social activities of patients with RLS, and question 3 was about the diagnostic criteria of RLS. The overall score indicated the RLS severity. A minimum score of 0 and a maximum score of 40 could be obtained. A score between 1 and 10 corresponded to "mild," 11-20 "moderate," 21-30 "severe," and 31-40 "very severe" RLS.
Kidney Disease Quality of Life Short Form (KDQOLTM-36) | change from baseline score at the end of one month
  This scale is used in determining the quality of life of HD patients and those who have end-stage renal disease (ESRD) stages 1-5. The Turkish validity and reliability study of the scale was conducted by Yıldırım et al., with a Cronbach's alpha value of 0.84-0.91. KDQOLTM-36 is a personalized scale that includes general tests supported by multi-question scales targeting specific problems such as symptoms, effects of kidney disease on daily life, burden of the kidney disease, working status, cognitive functions, quality of social relations, sexual functions, and sleep among dialysis patients with kidney disease. Patients are asked questions based on the past month. The total and subscale scores were calculated based on the KDQOLTM-36 scoring program. Each item was scored using Likert's method. The scores range from 0 to 100, and higher scores indicated better health-related quality of life. "0" indicated the worst health status, whereas "100" indicated the best health status.

CONTACTS AND LOCATIONS:
Overall Officials: AYSER DÖNER, Principal Investigator — TC Erciyes University
Locations (1):
- Department of Internal Nursing, Faculty of Health Science, Erciyes University, Kayseri, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans.

REFERENCES:
- [Result] Al-Jahdali HH, Al-Qadhi WA, Khogeer HA, Al-Hejaili FF, Al-Ghamdi SM, Al Sayyari AA. Restless legs syndrome in patients on dialysis. Saudi J Kidney Dis Transpl. 2009 May;20(3):378-85. PMID 19414938
- [Result] Giannaki CD, Hadjigavriel M, Lazarou A, Michael A, Damianou L, Atmatzidis E, Stefanidis I, Hadjigeorgiou GM, Sakkas GK, Pantzaris M. Restless legs syndrome is contributing to fatigue and low quality of life levels in hemodialysis patients. World J Nephrol. 2017 Sep 6;6(5):236-242. doi: 10.5527/wjn.v6.i5.236. PMID 28948161
- [Result] Kutlu R, Selcuk NY, Sayin S, Kal O. Restless legs syndrome and quality of life in chronic hemodialysis patients. Niger J Clin Pract. 2018 May;21(5):573-577. doi: 10.4103/njcp.njcp_84_17. PMID 29735856
- [Result] Lin XW, Zhang JF, Qiu MY, Ni LY, Yu HL, Kuo SH, Ondo WG, Yu Q, Wu YC. Restless legs syndrome in end stage renal disease patients undergoing hemodialysis. BMC Neurol. 2019 Mar 29;19(1):47. doi: 10.1186/s12883-019-1265-y. PMID 30925907
- [Result] Hashemi SH, Hajbagheri A, Aghajani M. The Effect of Massage With Lavender Oil on Restless Leg Syndrome in Hemodialysis Patients: A Randomized Controlled Trial. Nurs Midwifery Stud. 2015 Dec;4(4):e29617. doi: 10.17795/nmsjournal29617. Epub 2015 Dec 1. PMID 26835466
- [Result] Muz G, Tasci S. Effect of aromatherapy via inhalation on the sleep quality and fatigue level in people undergoing hemodialysis. Appl Nurs Res. 2017 Oct;37:28-35. doi: 10.1016/j.apnr.2017.07.004. Epub 2017 Aug 1. PMID 28985917
- [Result] Cevik B, Tasci S. The effect of acupressure on upper extremity pain and quality of life in patients hemodialysis treatment: A Randomized Controlled Trial. Complement Ther Clin Pract. 2020 May;39:101128. doi: 10.1016/j.ctcp.2020.101128. Epub 2020 Mar 2. PMID 32379666
- [Result] Allen RP, Picchietti D, Hening WA, Trenkwalder C, Walters AS, Montplaisi J; Restless Legs Syndrome Diagnosis and Epidemiology workshop at the National Institutes of Health; International Restless Legs Syndrome Study Group. Restless legs syndrome: diagnostic criteria, special considerations, and epidemiology. A report from the restless legs syndrome diagnosis and epidemiology workshop at the National Institutes of Health. Sleep Med. 2003 Mar;4(2):101-19. doi: 10.1016/s1389-9457(03)00010-8. PMID 14592341
- [Result] Allen RP, Picchietti DL, Garcia-Borreguero D, Ondo WG, Walters AS, Winkelman JW, Zucconi M, Ferri R, Trenkwalder C, Lee HB; International Restless Legs Syndrome Study Group. Restless legs syndrome/Willis-Ekbom disease diagnostic criteria: updated International Restless Legs Syndrome Study Group (IRLSSG) consensus criteria--history, rationale, description, and significance. Sleep Med. 2014 Aug;15(8):860-73. doi: 10.1016/j.sleep.2014.03.025. Epub 2014 May 17. PMID 25023924
- [Result] Hening WA, Allen RP. Restless legs syndrome (RLS): the continuing development of diagnostic standards and severity measures. Sleep Med. 2003 Mar;4(2):95-7. doi: 10.1016/s1389-9457(03)00009-1. No abstract available. PMID 14592339
- [Result] Walters AS, LeBrocq C, Dhar A, Hening W, Rosen R, Allen RP, Trenkwalder C; International Restless Legs Syndrome Study Group. Validation of the International Restless Legs Syndrome Study Group rating scale for restless legs syndrome. Sleep Med. 2003 Mar;4(2):121-32. doi: 10.1016/s1389-9457(02)00258-7. PMID 14592342
- [Result] Yildirim A, Ogutmen B, Bektas G, Isci E, Mete M, Tolgay HI. Translation, cultural adaptation, initial reliability, and validation of the Kidney Disease and Quality of Life-Short Form (KDQOL-SF 1.3) in Turkey. Transplant Proc. 2007 Jan-Feb;39(1):51-4. doi: 10.1016/j.transproceed.2006.10.196. PMID 17275473
- [Result] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Result] Mirbagher Ajorpaz N, Rahemi Z, Aghajani M, Hashemi SH. Effects of glycerin oil and lavender oil massages on hemodialysis patients' restless legs syndrome. J Bodyw Mov Ther. 2020 Jan;24(1):88-92. doi: 10.1016/j.jbmt.2019.06.012. Epub 2019 Jun 29. PMID 31987569
- [Result] Nasiri M, Abbasi M, Khosroabadi ZY, Saghafi H, Hamzeei F, Amiri MH, Yusefi H. Short-term effects of massage with olive oil on the severity of uremic restless legs syndrome: A double-blind placebo-controlled trial. Complement Ther Med. 2019 Jun;44:261-268. doi: 10.1016/j.ctim.2019.05.009. Epub 2019 May 8. PMID 31126564
- [Derived] Doner A, Tasci S. Effect of massage therapy with lavender oil on severity of restless legs syndrome and quality of life in hemodialysis patients. J Nurs Scholarsh. 2022 May;54(3):304-314. doi: 10.1111/jnu.12738. Epub 2021 Nov 14. PMID 34779137